CLINICAL TRIAL: NCT00929487
Title: Acute Clinical Evaluation of MPS in Soft Contact Lens Wearers
Brief Title: Acute Clinical Evaluation of Multi-purpose Solutions (MPS) in Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SMA-09-14/RDG-11-152
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Myopia
Keywords: contact lens wear; contact lens solution; corneal staining
MeSH Terms: conditions — Myopia | interventions — Sodium Chloride; Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Contact lens solution #1 (Experimental)
  Interventions: Device: Contact lens multi-purpose solution; Device: Contact lenses
- Contact lens solution #2 (Experimental)
  Interventions: Device: Contact lens multi-purpose solution; Device: Contact lenses
- Contact lens solution #3 (Experimental)
  Interventions: Device: Contact lens multi-purpose solution; Device: Contact lenses
- Contact lens solution #4 (Experimental)
  Interventions: Device: Contact lens multi-purpose solution; Device: Contact lenses
- Saline/blister pack solution (Active Comparator)
  Interventions: Other: Saline/blister pack solution; Device: Contact lenses

INTERVENTIONS:
Device: Contact lens multi-purpose solution — Lens care solutions CE-marked for intended use. A fresh pair of contact lenses was soaked overnight in the test contact lens solution and a pre-cycled lens case prior to study visit, then worn for two hours on the day of the study visit. Up to four solutions were evaluated in randomized order with the same brand of contact lenses, and a minimum of 12 hours of no lens wear separated each wear period.
  Other Names: ReNu Multiplus; Ote Hydroshield; Sauflon Synergi; Lapis Lazuli Eye See Aqua Balance; Avizor All Clean Soft; Sauflon Cyclean; Vita Research Regard; Menicon MeniCare Soft; ALL; ReNu MPS; Welcon; Hydron
  Arms: Contact lens solution #1; Contact lens solution #2; Contact lens solution #3; Contact lens solution #4
Other: Saline/blister pack solution — A fresh pair of contact lenses was soaked overnight in saline prior to study visit or was inserted directly from the blister pack, then worn for two hours on the day of the study visit.
  Other Names: AMO OcuPure Saline; Saline
  Arms: Saline/blister pack solution
Device: Contact lenses — CE-marked silicone hydrogel contact lenses soaked overnight for at least 10 hours prior to the study visit, then worn for two hours on the day of the study visit. A fresh pair of the same brand of contact lenses was used for each overnight soak (ie, 4 solutions plus saline/blister pack solution), and a minimum of 12 hours separated each wear period.
  Other Names: PureVision; Air Optix Aqua; Acuvue Advance; Biofinity

SUMMARY:
The purpose of this study was to clinically evaluate lens care solutions used with soft contact lenses.

DETAILED DESCRIPTION:
This study was conducted as a series of ten smaller studies in three countries using commercially available contact lens solutions per each country, ie, United Kingdom, France, and the Philippines. In each study, participants were assessed after use of up to 5 products (with one always being a control saline/blister pack solution) in randomized order in conjunction with one of the silicone hydrogel contact lenses. A total of 278 participants were enrolled in the 10 studies.

ELIGIBILITY:
Inclusion Criteria:

* Have read, understood, signed, and dated the written Informed Consent.
* Be an adapted and successful soft contact lens wearer on a daily wear basis for at least two weeks.
* Vision correctable to at least 20/30 Snellen.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Topical ocular medication use.
* History of hypersensitivity to any component of the study contact lens care systems.
* Any slit-lamp finding of abnormal nature at the baseline visit assessment of each study period.
* Pregnant, lactating, or planning a pregnancy.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Corneal Staining | 2 hours

SECONDARY OUTCOMES:
Subjective Comfort | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Visioncare Research, Ltd., Farnham, Surrey, United Kingdom

REFERENCES:
- [Derived] Malet F. An acute clinical comparison of corneal staining and comfort associated with contact lens care solutions. Cont Lens Anterior Eye. 2014 Oct;37(5):351-7. doi: 10.1016/j.clae.2014.05.007. Epub 2014 Jul 26. PMID 25070393